CLINICAL TRIAL: NCT03259464
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 685509 in Healthy Chinese and Japanese Male Volunteers (Randomised, Single-blind, Placebo-controlled Trial)
Brief Title: This Study Tests BI 685509 in Healthy Chinese and Japanese Men; the Study Tests How Different Doses of BI 685509 Are Taken up in the Body and How Well They Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1366-0013
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 685509 (Experimental): Chinese & Japanese subjects
  Interventions: Drug: BI 685509
- Placebo (Placebo Comparator): Chinese & Japanese subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 685509 — 3 sequential dose groups
  Arms: BI 685509
Drug: Placebo — 3 sequential dose groups
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 685509 in healthy male subjects following oral administration of multiple rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) and pharmacodynamics (PD) of BI 685509 in healthy Chinese and Japanese subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Chinese or Japanese ethnicity, according to the following criteria:

  * Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
  * Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years (incl.)
* Body mass index (BMI) range: ≥18.5 and <25.0 kg/m2
* Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation.
* Male subjects who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 90 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: combined oral contraceptives, intrauterine device
  * Vasectomised (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy) female partner
  * Sexually abstinent

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including HIV, viral hepatitis and (or) tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold (or TSPOT) test. Subjects with a positive QuantiFERON TB-Gold (or T-SPOT) test will not participate in the study. The HBV carriers and subjects with history of HB (including the subjects with only HBs antibody positive [negative for both HBs antigen and HBc antibody] and without HB vaccination) will not be allowed to participate in this trial.
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of biologic agents other than current study medication or drugs considered likely to interfere with the safe conduct of the study
* Within 30 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial (including bioequivalence trial) with an investigational drug within 90 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 200 mL within 30 days or 400 mL within 12 weeks prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Have received any live bacterial or live viral vaccination in the 12 weeks prior to the date of screening. Subjects must agree not to receive a live bacterial or live viral vaccination during the study and up to 12 months after the last administration of study drug
* Have received Bacille Calmette-Guerin (BCG) vaccination in the 12 months prior to the date of screening. Subjects must agree not to receive BCG vaccination during the study and up to 12 months after the last administration of study drug
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-05-26 (Actual)

PRIMARY OUTCOMES:
Number [N (%)] of subjects with drug-related Adverse Events (AEs) | up to day 35

SECONDARY OUTCOMES:
After the first dose:AUC0-24 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h) | up to 24 hours
After the first dose:Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours
After the drug administration on Day 10 and Day 17 of DGs 1-2: AUCtau,ss (area under the concentration-time curve of the analyte in plasma over the dosing interval tau at steady state) [AUCtau,ss will be AUC0-12,ss for b.i.d. and AUC0-24,ss for q.d.] | Dose Group (DG) 1: up to 240 hours & up to 408 hours DG2: up to 240 hours & up to 396 hours
After the drug administration on Day 10 and Day 17 of DGs 1-2: Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) | Dose Group (DG) 1: up to 240 hours & up to 408 hours DG2: up to 240 hours & up to 396 hours

CONTACTS AND LOCATIONS:
Locations (2):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan
- Seoul National University Hospital, Seoul, South Korea